CLINICAL TRIAL: NCT02745288
Title: Inferior Alveolar Nerve Block for Intraoperative Analgesia for Maxillofacial Cancer Surgery Requiring Unilateral Mandibular Resection-A Randomized Controlled Study
Brief Title: Inferior Alveolar Nerve Block for Intraoperative Analgesia for Maxillofacial Cancer Surgery - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Madhavi Shetmahajan, Associate professor, dept of anaethesia, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1648
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Mandibular Neoplasms
MeSH Terms: conditions — Mandibular Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve block (Experimental): This arm will receive inferior alveolar nerve block
  Interventions: Procedure: inferior alveolar nerve block
- control (No Intervention): Control arm will not receive inferior alveolar block

INTERVENTIONS:
Procedure: inferior alveolar nerve block — A long acting local anaesthetic agent Inj Bupivacaine hydrochloride 0.5% (2 ml) will be given after induction by open mouth technique by landmark method.
  The mucobuccal fold will be palpated and traced till coronoid notch. The finger will be moved medially across the retromandibular trigone on internal oblique ridge. The 25G needle will be inserted till bone is felt. 2 ml of 0.5% bupivacaine will be injected slowly after withdrawing needle by 1mm and confirming negative aspiration of blood.
  Arms: Nerve block

SUMMARY:
Mandibular resection which is an important component of maxillofacial cancer surgery is an extremely painful procedure associated with severe sympathetic response needing high doses of opioids. Inferior alveolar nerve block is a common nerve block used by dentists for mandibular dental extractions. The aim of this trial is to study the effect of this block for intraoperative analgesia in maxillofacial cancer surgeries requiring unilateral mandibular resection.

DETAILED DESCRIPTION:
All adult patients below 75yrs of age scheduled for maxillofacial surgery will be screened for inclusion and exclusion criteria.

Written informed consent will be taken one day prior to surgery. Consenting subjects will be randomized after induction of anaesthesia to study or control arm.

The duration of the study is from induction of anaesthesia to the completion of primary tumour removal and neck dissection

Study procedure: Ipsilateral Inferior alveolar nerve block A long acting local anaesthetic agent Inj Bupivacaine hydrochloride 0.5% (2 ml) will be given after induction by open mouth technique by landmark method.

The mucobuccal fold will be palpated and traced till coronoid notch. The finger will be moved medially across the retromandibular trigone on internal oblique ridge. The 25G needle will be inserted till bone is felt. 2 ml of 0.5% bupivacaine will be injected slowly after withdrawing needle by 1mm and confirming negative aspiration of blood.

Control arm will not receive any intervention. The study investigator will give a mock injection for blinding of the attending anaesthetist

The study procedure will be done by the study investigators 10 -30 minutes prior to commencing surgery for primary tumour.

Account of procedure:

All patients will have standard conduct of anaesthesia except for the alveolar nerve injection in the study group.

All patients will have the minimum standard monitoring of pulse oximeter, electrocardiogram, capnography and non invasive blood pressure monitoring.

Blood pressure and heart rate will be recorded every 5 min interval from the beginning till completion of primary tumor excision and neck dissection

Induction of anaesthesia: IV fentanyl 2 mcg/kg, IV Propofol 2 -3 mg/kg. IV neuromuscular blocking agent used will be Inj vecuronium bromide in the dose of 0.1 mg /kg. All patients will have standard airway management at the discretion of the attending anaesthesiologist.

Intraoperative maintenance of anaesthesia will be as follows

1. Controlled ventilation with isoflurane in air / oxygen with minimal alveolar concentration of 0.8 -1.2
2. Intraoperative analgesic - IV fentanyl in boluses of 1 mcg/kg at the discretion of the anaesthetist based on the haemodynamic response till the completion of primary tumour removal and neck dissection. Thereafter, the choice of analgesic will be left to the anaesthetist
3. In case of uncontrolled sympathetic response (hypertension and/or tachycardia) to surgery not controlled by IV fentanyl (10 mcg/kg ), rescue intraoperative analgesic/ anaesthetic (e.g.IV morphine, IV diclofenac, IV dexmedetomide, IV propofol, increase in inhalational anaesthetic concentration, etc) or vasoactive agents (e.g.IV Esmolol, IV Nitroglycerin, etc) may be used. This will be noted in the Case record form.

Information will be collected as per Case Record form by the investigator. Any deviation from protocol will be recorded.

Sample size calculation Based on the average fentanyl requirement 340mcg found in pilot data, to detect 25% reduction in fentanyl requirement in the study group compared to control group, with 80% power and level of significance of 5% ,the sample size calculated was 22 in each group.

Statistical Analysis The fentanyl requirement in the two groups, maximum heart rate and maximum blood pressure will be will be compared using students t test Other variables will be described as numbers and percentage

Demographic ,clinical and disease relate variable will be present as frequency (percentage) and mean (S.D.) or median as appropriate.

Two group comparisons will be made using independent t-test or Man Whitney U test as per distribution of the data.

P-value< 0.05 will be considered statistical significant. Repeated measures ANOVA will be used to compare change of blood pressure and heart rate from baseline at various time points.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the age of 18 and 75 yrs classified as ASA I and II physical status requiring maxillofacial cancer surgery requiring unilateral mandibular resection and unilateral neck dissection

Exclusion Criteria:

* - surgery involving upper alveolar / maxillary resection
* patients with BMI below 18kg/m2 and above 30kg/m2
* allergy to local anaesthetic agent
* Inability to give inferior alveolar nerve block due to any cause e.g. restricted mouth opening, obscured landmark or infection at site
* pregnant women
* patients unable to give valid consent e.g. patients with learning difficulties
* patients on medications for hypertension
* patients with preoperative pain requiring regular pain medications
* uncontrolled haemodynamic status e.g. baseline arterial blood pressure above 160 /90 and baseline HR above 100 /min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
IV fentanyl requirement during primary tumour removal | From start to finish ofprimary tumour removal procedure
  The total IV fentanyl dose required during primary tumour removal will be noted

SECONDARY OUTCOMES:
IV fentanyl requirement during neck dissection and primary tumour removal | From start to finish of neck dissection and primary tumour removal
  The total IV fentanyl dose required during neck dissection and primary tumour removal will be noted
Maximum change in heart rate from baseline during primary tumour removal | From start to finish of primary tumour removal procedure
Maximum change in blood pressure from baseline during primary tumour removal | From start to finish of primary tumour removal procedure
Need for rescue analgesics or vasoactive agents during primary tumour removal | From start to finish of primary tumour removal procedure

CONTACTS AND LOCATIONS:
Overall Officials: Madhavi Shetmahajan, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, India, India

IPD SHARING:
Plan to Share IPD: No